CLINICAL TRIAL: NCT02919930
Title: Interface Selection for Adaptive Servo Ventilation: A Randomized Controlled Study
Brief Title: Interface Selection for Adaptive Servo Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S57607
Record Dates: First submitted 2016-06-30; First posted 2016-09-30 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Central Sleep Apnea; ASV
MeSH Terms: conditions — Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oronasal - Nasal (Other): Patients undergo polysomnography with oronasal mask during the first night and nasal mask during the second night.
  Interventions: Device: Switch from oronasal to nasal mask during ASV treatment
- Nasal - Oronasal (Other): Patients undergo polysomnography with nasal mask during the first night and oronasal mask during the second night.
  Interventions: Device: Switch from nasal to oronasal mask during ASV treatment

INTERVENTIONS:
Device: Switch from oronasal to nasal mask during ASV treatment — One night of ASV treatment with oronasal mask followed by one night of ASV treatment with nasal mask.
  Arms: Oronasal - Nasal
Device: Switch from nasal to oronasal mask during ASV treatment — One night of ASV treatment with nasal mask followed by one night of ASV treatment with oronasal mask.
  Arms: Nasal - Oronasal

SUMMARY:
The purpose of this study is to compare the effects of nasal and oronasal interfaces during ASV treatment on sleep efficiency and sleep architecture. Therefore, patients starting treatment with ASV, will be randomized between two groups. In the first group, patients will use a nasal interface during the first night and an oronasal interface during the second night. In the second group, patients will use an oronasal mask first and a nasal mask during the second night. The results of this trial will have major impact on future clinical practice as it would deliver prediction rules to choose the correct interface immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patients with central sleep apnea, not responding to treatment with CPAP
* Indication for treatment with ASV

Exclusion Criteria:

* Patients < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Apnea/hypopnea index | Two nights
  Effect on respiratory events

SECONDARY OUTCOMES:
Mask comfort VAS | Two nights
  Subjective mask comfort
Device leaks data | Two nights
  Evaluation of leaks (data of ASV device)
Sleep efficiency | Two nights
  polysomnographic evaluation
Sleep architecture | Two nights
  Polysomnographic evaluation of different sleep stages

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No